CLINICAL TRIAL: NCT00462735
Title: Phase II Study of Concomitant Fluorouracil, Hydroxyurea, Cetuximab and Hyperfractionated Intensity Modulated Radiation Therapy for Locally Advanced Head and Neck Cancer
Brief Title: Fluorouracil, Hydroxyurea, Cetuximab and Twice-daily Intensity Radiation Therapy for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnny Kao (Other)
Responsible Party: Sponsor-Investigator, Johnny Kao, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 06-1155
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Head and Neck Cancer; Cancer of the Pharynx; Cancer of the Larynx; Nose Neoplasms; Paranasal Sinus Neoplasms; Cancer of the Oral Cavity
Keywords: Cancer of the Nasal Cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Pharyngeal Neoplasms; Laryngeal Neoplasms; Nose Neoplasms; Paranasal Sinus Neoplasms | interventions — Cetuximab; Hydroxyurea; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Advanced Head and Neck Cancer (Experimental): Patients with stage IVA and IVB or high-risk stage III squamous cell carcinomas of the head and neck
  Interventions: Drug: Cetuximab; Drug: Hydroxyurea; Drug: Fluorouracil; Procedure: radiotherapy

INTERVENTIONS:
Drug: Cetuximab — 250 mg/m2 on Day 1 after the first dose of radiation was administered to all patients
Drug: Hydroxyurea — 500 mg orally every 12 hours with the morning dose administered 2 hours before radiation
Drug: Fluorouracil — continuous-infusion 5-FU at a dose of 600 mg/m2 daily for 120 hours
Procedure: radiotherapy — Radiotherapy was administered at 1.5 Gy per fraction twice daily with treatments separated by at least 6 hours on Days 1 through 5 on an alternating week schedule.
  Radiation was delivered with intensity-modulated radiation therapy (IMRT) planning for all patients.

SUMMARY:
For advanced head and neck cancer, combined radiation and chemotherapy prevents recurrences and for many patients, improves survival. While combined cisplatin and radiation or cetuximab and radiation is more effective than radiation alone, approximately 50% of these patients will still recur. A more aggressive approach may be needed for these patients to prevent recurrence and death. The strategy of using multiple chemotherapy drugs with radiation given twice a day has been tested at Mount Sinai and University of Chicago. Approximately 80% of patients are cured with this strategy. While cure rates are higher than standard chemotherapy and radiation and the treatment is tolerable, side effects during treatment are common. We propose replacing a chemotherapy drug with a less toxic, targeted therapy called cetuximab. Our goal is to reduce toxicity while maintaining or improving cure rates for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas of the head and neck or lymphoepithelioma
* No prior chemotherapy or radiotherapy
* Prior surgical therapy will consist only of incisional or excisional biopsy, and organ sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an existing primary tumor
* Karnofsky performance status of >= 70%
* Intact organ and bone marrow function
* Obtained informed consent

Exclusion Criteria:

* Demonstration of metastatic disease (i.e. M1 disease).
* Patients with a history of severe allergic reaction to docetaxel or other drugs formulated with polysorbate 80. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, 5-fluorouracil, or hydroxyurea.
* Other coexisting malignancies or malignancies diagnosed within the previous 3 years with the exception of basal cell carcinoma, cervical cancer in situ, and other treated malignancies with no evidence of disease for at least 3 years.
* Prior surgical therapy other than incisional or excisional biopsy and organ-sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an unknown primary tumor. Any non-biopsy procedure must have taken place less than 3 months from initiating protocol treatment.
* Incomplete healing from previous surgery
* Pregnancy or breast feeding (men and women of child-bearing potential are eligible but must consent to using effective contraception during therapy and for at least 3 months after completing therapy)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary artery disease will be at the discretion of the attending physician.
* Uncontrolled active infection unless curable with treatment of their cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Kao, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Kao J, Genden EM, Gupta V, Policarpio EL, Burri RJ, Rivera M, Gurudutt V, Som PM, Teng M, Packer SH. Phase 2 trial of concurrent 5-fluorouracil, hydroxyurea, cetuximab, and hyperfractionated intensity-modulated radiation therapy for locally advanced head and neck cancer. Cancer. 2011 Jan 15;117(2):318-26. doi: 10.1002/cncr.25374. Epub 2010 Sep 9. PMID 20830768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period January 2007 through April 2008. All cases were reviewed at a multidisciplinary conference, which was attended by representatives from the Departments of Head and Neck Surgery, Radiation Oncology, Medical Oncology, Palliative Care, Social Work, and Nutrition at Icahn School of Medicine at Mount Sinai.
Groups:
- Advanced Head and Neck Cancer: Patients with stage IVA and IVB or high-risk stage III squamous cell carcinomas of the head and neck. Cetuximab- 250 mg/m2 on Day 1 after the first dose of radiation was administered to all patients. Hydroxyurea - 500 mg orally every 12 hours with the morning dose administered 2 hours before radiation. Fluorouracil - continuous-infusion 5-FU at a dose of 600 mg/m2 daily for 120 hours. Radiotherapy.
  Radiotherapy was administered at 1.5 Gy per fraction twice daily with treatments separated by at least 6 hours on Days 1 through 5 on an alternating week schedule.
  Radiation was delivered with intensity-modulated radiation therapy (IMRT) planning for all patients.
Period: Overall Study
Arm/Group | Advanced Head and Neck Cancer
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Advanced Head and Neck Cancer: Cetuximab- 250 mg/m2 on Day 1 after the first dose of radiation was administered to all patients. Hydroxyurea - 500 mg orally every 12 hours with the morning dose administered 2 hours before radiation. Fluorouracil - continuous-infusion 5-FU at a dose of 600 mg/m2 daily for 120 hours. Radiotherapy.
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 59 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23
  Black | 5
  Hispanic | 5
  Asian | 0
Performance score [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG)
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2- Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  participants
    0 | 12
    1 | 19
    2 | 2
Charlson comorbidity score [Number; unit: participants] — The Charlson Comorbidity Index contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions. Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. Scores are summed to provide a total score to predict mortality. Higher scores indicating greater comorbidity (patients with a score > 5 have essentially a 100% risk of dying at one year).
  participants
    0-1 | 27
    ≥2 | 6
Alcohol consumption [Number; unit: participants]
  None | 10
  Occasional | 14
  Moderate | 2
  Heavy | 7
Smoking [Number; unit: participants]
  None | 6
  Cigar, pipe, or betel nut only | 3
  ≤20 pack-y | 9
  20.1-40 packk-y | 7
  >40 pack-y | 8
Primary site [Number; unit: participants]
  Sinonasal | 2
  Nasopharynx | 2
  Oropharynx | 14
  Oral cavity | 6
  Salivary gland | 1
  Larynx | 2
  Hyopharynx | 4
  Unknown primary | 2

OUTCOME MEASURES:

1. Primary Outcome: Llocoregional Recurrence
Description: Percentage of Participants with Loco-regional recurrence.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 33
Participants | 27

2. Primary Outcome: Survival
Description: Overall Survival - Percentage of Participants who survived Disease-Free Survival - measured from the initiation of nonsurgical treatment to either the last follow-up, disease progression, or death using intent-to-treat methodology
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 33
percentage of participants
  Overall Survival | 86
  Disease-Free Survival | 69

3. Secondary Outcome: Long- Term Toxicity
Description: Grade 3 toxicities events
Time Frame: 2 years
Measure: Number; unit: events
Groups:
- Advanced Head and Neck Cancer: Cetuximab - 250 mg/m2 on Day 1 after the first dose of radiation was administered to all patients. Hydroxyurea - 500 mg orally every 12 hours with the morning dose administered 2 hours before radiation. Fluorouracil - continuous-infusion 5-FU at a dose of 600 mg/m2 daily for 120 hours. Radiotherapy.
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 33
events | 32

4. Secondary Outcome: UW-QOLR: Quality of Life Score
Description: University of Washington Quality of Life (UW-QOLR) questionnaire - covers 12 domains - pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder function, taste, saliva, mood and anxiety. Each domain have between 3 and 6 response options that are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response and reported as one composite score from 0 (worst) to 100 (best).
Time Frame: 2 years
Population: Twenty patients completed the UW-QOLR questionnaire before and after therapy.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 20
units on a scale | 80 [0 to 100]

5. Secondary Outcome: Distant Metastases
Description: Percentage of participants who did not have distant control
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Advanced Head and Neck Cancer
Number analyzed (Participants) | 33
percentage of participants | 21

ADVERSE EVENTS:
Arm/Group | Advanced Head and Neck Cancer
Serious Adverse Events (participants affected / at risk) | 33/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Head and Neck Cancer (N=33)
Mucositis (Gastrointestinal disorders) | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Pain (General disorders) | 14
Low Absolute neutrophil count (Blood and lymphatic system disorders) | 4
Low White blood count (Blood and lymphatic system disorders) | 6
Low Hemoglobin count (Blood and lymphatic system disorders) | 6
Low Platelets count (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Head and Neck Cancer (N=33)
Mucositis (Gastrointestinal disorders) | 22
Dermatitis (Skin and subcutaneous tissue disorders) | 28
Pain (General disorders) | 19
Xerostomia (General disorders) | 33
Low Absolute neutrophil count (Blood and lymphatic system disorders) | 18
Low White blood count (Blood and lymphatic system disorders) | 25
Low Hemoglobin count (Blood and lymphatic system disorders) | 25
Low Platelet count (Blood and lymphatic system disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes